CLINICAL TRIAL: NCT05399550
Title: A Phase II, Randomized, Double Blind, Placebo Controlled Multicenter Study to Evaluate The Safety and Efficacy of Balovaptan in Patients With Acute Ischemic Stroke at High Risk of Developing Malignant Cerebral Edema
Brief Title: Study to Evaluate The Safety and Efficacy of Balovaptan in Participants With Acute Ischemic Stroke at a High Risk of Developing Malignant Brain Edema
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WC 42759
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — balovaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Balovaptan (Experimental): Balovaptan will be administered as IV infusion once a day over 3 days
  Interventions: Drug: Balovaptan
- Placebo (Placebo Comparator): Placebo will be administered as IV infusion once a day over 3 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Balovaptan — Intravenous Solution
  Arms: Balovaptan
Drug: Placebo — Matching Intravenous Solution
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the safety, efficacy, and pharmacokinetics of balovaptan compared with placebo in participants with acute ischemic stroke (AIS) at risk of developing Malignant Cerebral Edema (MCE)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of LVO in the anterior circulation such that study drug administration can be initiated within 12 hours of LKW and at risk of MCE development, as defined as follows:
* Documented occlusion of terminus ICA and/or MCA on CTA or magnetic resonance angiogram and
* ASPECTS score </=5 on NCCT and
* NIHSS >15 for the non-dominant hemisphere and >20 for the dominant hemisphere (or > 20 if dominant/non-dominant hemisphere unknown)
* Present with a WUS </=8 hours from awakening provided the above criteria are met
* Participants with a history of seizures on anti-epileptic medications may be included if they have been on stable doses of those medications for at least 12 weeks prior to LKW, they have not experienced seizures during that time frame, and their anti-epileptic medicines are continued during the study
* For women of childbearing potential: participants who agree to remain abstinent (refrain from heterosexual intercourse) or use contraception and agree to refrain from donating eggs
* No specific contraception methods for males are required.

Exclusion Criteria:

* Participants who are >12 hours from LKW at the start of treatment with study drug or >8 hours from awakening with WUS
* Any MLS on brain imaging
* Evidence of intracranial hemorrhage at screening based on NCCT
* Contraindication to MRI examination
* Evidence of additional anterior cerebral artery (ACA) infarction
* Diagnosis of brain death
* Planned surgical decompression prior to randomization
* Participants with a known history of a hereditary bleeding disorder which increases bleeding risk
* Chronic kidney disease stage III or higher
* Hepatic injury
* Diagnosis of diabetes insipidus
* Participants who have received any prophylactic hyperosmolar therapy
* Participants who have received treatment with any other V1a and/or V2 receptor-blocking agent or glyburide
* A preexisting medical condition for which the participant is unlikely to survive the next 6 months
* Planned limitation or withdrawal of life-sustaining treatment during hospital admission
* Participants who are pregnant or breastfeeding, or intending to become pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Amount of midline shift (MLS) at 72 hours from Last Known Well (LKW) | 72 Hours from Last Known Well
  Midline shift will be measured in millimeter on non-contrast computer tomography (NCCT)

SECONDARY OUTCOMES:
Percentage of Participants with modified Rankin Scale-Structured Interview (mRS-SI) score </= 4 vs. >4 | At Day 90
Amount of MLS | At 48 hours and 96-120 hours from LKW
  MLS will be measured in millimeter on NCCT
Percentage of Participants with Surgical DHC Performed | From Baseline up to Day 90
Percentage of Participants Who Received Hyperosmolar therapy following initiation of study treatment | From Baseline up to Day 90
National Institute of Health Stroke Scale (NIHSS) score | At Day 4 and Day 90
Mortality | At Day 30
  Mortality in the first 30 days after the enrollment
mRS-SI score | At Day 30
Functional Independence Measure (FIM) score | At Discharge or Day 10 and Day 90
Glasgow Outcome Scale Extended (GOSE) Score | at Discharge or Day 10, Day 30 and Day 90
Stroke Impact Scale-16 (SIS-16) score | At Day 30 and Day 90
Length (in days) of ICU and Hospital Stay | From Baseline to Day 90
Number of participants with adverse events and severity of adverse events | From Baseline to Day 90
  Severity will be determined according to the NCI CTCAE v5.0
Plasma concentrations of balovaptan at specified timepoints | From Baseline to 120 Hours After the End of the Last Infusion (or at discharge)
Area under the concentration-time curve from Time 0 to 24 hours after a given dose (AUC24hr) | From Baseline to 120 Hours After the End of the Last Infusion (or at discharge)]
  As calculated by NCA from measured concentration
Maximum observed concentration (Cmax) | From Baseline to 120 Hours After the End of the Last Infusion (or at discharge)]
  As calculated by NCA or taken directly from measured concentration
Plasma drug concentration 24hours after the administration of a given dose (C24hr) | From Baseline to 120 Hours After the End of the Last Infusion (or at discharge)]
  As calculated by NCA or taken directly from measured concentration
Number of participants with safety findings on brain imaging | From Baseline to Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- CPMC Comprehensive Stroke Care Center, San Francisco, California, United States